CLINICAL TRIAL: NCT02185794
Title: Phase 1b, Randomized, Double-Blind, Multiple-Dose Ranging Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of GS-9857 in Subjects With Chronic Hepatitis C Virus Infection
Brief Title: Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of Voxilaprevir in Adults With Chronic Hepatitis C Virus Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-338-1121
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-08

CONDITIONS: Hepatitis C Virus Infection
Keywords: Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; Enterovirus Infections; Picornaviridae Infections; RNA Virus Infections; Flaviviridae Infections; Antiviral Agents; Anti-Infective Agents; Therapeutic Uses; Pharmacologic Actions; Antimetabolites; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Hepatitis C; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; Enterovirus Infections; Picornaviridae Infections; RNA Virus Infections; Flaviviridae Infections | interventions — voxilaprevir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- Placebo (GT 1a, Cohort 1) (Placebo Comparator): Participants with genotype (GT) 1a HCV infection will receive placebo once daily for 3 days under fasted conditions.
  Interventions: Drug: Placebo to match voxilaprevir
- Voxilaprevir 50 mg (GT 1a, Cohort 1) (Experimental): Participants with GT 1a HCV infection will receive voxilaprevir 50 mg once daily for 3 days under fasted conditions.
  Interventions: Drug: Voxilaprevir
- Voxilaprevir 100 mg (GT 1a, Cohort 1) (Experimental): Participants with GT 1a HCV infection will receive voxilaprevir 100 mg once daily for 3 days under fasted conditions.
  Interventions: Drug: Voxilaprevir
- Voxilaprevir 300 mg (GT 1a, Cohort 1) (Experimental): Participants with GT 1a HCV infection will receive voxilaprevir 300 mg once daily for 3 days under fasted conditions.
  Interventions: Drug: Voxilaprevir
- Placebo (GT 3, Cohort 2) (Placebo Comparator): Participants with GT 3 HCV infection will receive placebo once daily for 3 days under fasted conditions.
  Interventions: Drug: Placebo to match voxilaprevir
- Voxilaprevir 50 mg (GT 3, Cohort 2) (Experimental): Participants with GT 3 HCV infection will receive voxilaprevir 50 mg once daily for 3 days under fasted conditions.
  Interventions: Drug: Voxilaprevir
- Voxilaprevir 100 mg (GT 3, Cohort 2) (Experimental): Participants with GT 3 HCV infection will receive voxilaprevir 100 mg once daily for 3 days under fasted conditions.
  Interventions: Drug: Voxilaprevir
- Voxilaprevir 300 mg (GT 3, Cohort 2) (Experimental): Participants with GT 3 HCV infection will receive voxilaprevir 300 mg once daily for 3 days under fasted conditions.
  Interventions: Drug: Voxilaprevir
- Placebo (GT 2, Cohort 3) (Placebo Comparator): Participants with GT 2 HCV infection will receive placebo once daily for 3 days under fasted conditions.
  Interventions: Drug: Placebo to match voxilaprevir
- Voxilaprevir 100 mg (GT 2, Cohort 3) (Experimental): Participants with GT 2 HCV infection will receive voxilaprevir 100 mg once daily for 3 days under fasted conditions.
  Interventions: Drug: Voxilaprevir
- Voxilaprevir 100 mg (GT 4, Cohort 4) (Experimental): Participants with GT 4 HCV infection will receive voxilaprevir 100 mg once daily for 3 days under fasted conditions.
  Interventions: Drug: Voxilaprevir
- Voxilaprevir 100 mg (GT 1b, Cohort 5) (Experimental): Participants with GT 1b HCV infection will receive voxilaprevir 100 mg once daily for 3 days under fasted conditions.
  Interventions: Drug: Voxilaprevir
- Voxilaprevir 100 mg Fed (GT 3a, Cohort 6) (Experimental): Participants with GT 3a HCV infection will receive voxilaprevir 100 mg once daily for 3 days under fed conditions.
  Interventions: Drug: Voxilaprevir
- Voxilaprevir 600 mg (Cohorts 7-9) (Experimental): Participants with genotypes 1a, 1b, 2, 3, or 4 HCV infection will receive voxilaprevir up to 600 mg under fasted or fed conditions for 3 days.
  Interventions: Drug: Voxilaprevir
- Voxilaprevir 100 mg + SOF/VEL 400/100 mg (Group 1, Cohort 10) (Experimental): Participants with any GT HCV infection received voxilaprevir 100 mg on Day 1 after moderate fat meal and voxilaprevir 100 mg plus sofosbuvir (SOF)/velpatasvir (VEL) (400/100 mg) fixed-dose combination (FDC)on Days 2 and 3 after either a light or moderate-fat meal.
  Interventions: Drug: Voxilaprevir; Drug: SOF/VEL
- Voxilaprevir 100 mg + SOF/VEL 400/100 mg (Group 2, Cohort 10) (Experimental): Participants with any GT HCV infection received voxilaprevir 100 mg on Day 1 and voxilaprevir 100 mg plus SOF/VEL (400/100 mg) FDC on Days 2 and 3 after moderate fat meal.
  Interventions: Drug: Voxilaprevir; Drug: SOF/VEL

INTERVENTIONS:
Drug: Voxilaprevir — Voxilaprevir tablets administered orally once daily
  Other Names: GS-9857
  Arms: Voxilaprevir 100 mg (GT 1a, Cohort 1); Voxilaprevir 100 mg (GT 1b, Cohort 5); Voxilaprevir 100 mg (GT 2, Cohort 3); Voxilaprevir 100 mg (GT 3, Cohort 2); Voxilaprevir 100 mg (GT 4, Cohort 4); Voxilaprevir 100 mg + SOF/VEL 400/100 mg (Group 1, Cohort 10); Voxilaprevir 100 mg + SOF/VEL 400/100 mg (Group 2, Cohort 10); Voxilaprevir 100 mg Fed (GT 3a, Cohort 6); Voxilaprevir 300 mg (GT 1a, Cohort 1); Voxilaprevir 300 mg (GT 3, Cohort 2); Voxilaprevir 50 mg (GT 1a, Cohort 1); Voxilaprevir 50 mg (GT 3, Cohort 2); Voxilaprevir 600 mg (Cohorts 7-9)
Drug: Placebo to match voxilaprevir — Placebo to match voxilaprevir tablets administered orally once daily
  Arms: Placebo (GT 1a, Cohort 1); Placebo (GT 2, Cohort 3); Placebo (GT 3, Cohort 2)
Drug: SOF/VEL — 400 mg/100 mg FDC tablet administered orally once daily
  Arms: Voxilaprevir 100 mg + SOF/VEL 400/100 mg (Group 1, Cohort 10); Voxilaprevir 100 mg + SOF/VEL 400/100 mg (Group 2, Cohort 10)

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of voxilaprevir (formerly GS-9857) alone or with sofosbuvir (SOF)/velpatasvir (VEL) fixed dose combination (FDC) and antiviral activity of voxilaprevir in adults with genotype 1, 2, 3, 4 hepatitis C virus (HCV) infection. All participants will be monitored for up to 48 weeks after the last dose.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic genotype 1-4 HCV infection
* For Cohorts 1-9, HCV RNA ≥ 100,000 IU/mL at screening (no HCV RNA restriction for Cohort 10)
* Screening laboratory values within defined thresholds
* Use of two effective contraception methods if female of childbearing potential or sexually active male

Key Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner
* Presence of cirrhosis
* Prior exposure to approved or experimental HCV Protease Inhibitors
* Co-infection with HIV or hepatitis B virus (HBV)
* Current or prior history of clinical hepatic decompensation
* Chronic use of systemic immunosuppressive agents
* History of clinically significant illness or any other medical disorder that may interfere with participant's treatment, assessment or compliance with the protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-06-13 (Actual); Primary Completion 2014-12-22 (Actual); Study Completion 2015-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (11):
- United States (10):
  - Costa Mesa, California
  - DeLand, Florida
  - Orlando, Florida
  - Kansas City, Missouri
  - St Louis, Missouri
  - Berlin, New Jersey
  - Marlton, New Jersey
  - Philadelphia, Pennsylvania
  - Knoxville, Tennessee
  - San Antonio, Texas
- San Juan, Puerto Rico

REFERENCES:
- [Result] Rodriguez-Torres M, Glass S, Hill J, Freilich B, Hassman D, Di Bisceglie A, Taylor J, Kirby B, Yang J, An D, Stamm L, Brainard D, Kim S, Krefetz D, Smith W, Marbury T, Lawitz E. The Pangenotypic NS3/4A Protease Inhibitor GS-9857 Demonstrates Potent Antiviral Activity in Patients Infected With HCV Genotype 1, 2, 3, or 4 in a 3-Day Monotherapy Study [Poster P0901]. Presented at the European Association for the Study of the Liver (EASL) 50th International Liver Congress 2015, April 22-26, 2015, Vienna, Austria.
- [Result] Lawitz E, Yang JC, Stamm LM, Taylor JG, Cheng G, Brainard DM, Miller MD, Mo H, Dvory-Sobol H. Characterization of HCV resistance from a 3-day monotherapy study of voxilaprevir, a novel pangenotypic NS3/4A protease inhibitor. Antivir Ther. 2018;23(4):325-334. doi: 10.3851/IMP3202. PMID 29063860

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States and Puerto Rico. The first participant was screened on 13 June 2014. The last study visit occurred on 28 September 2015.
Pre-assignment Details: Participants were enrolled in Cohorts 1, 2, 3, 4, 5, 6 and 10. Cohorts 7, 8, and 9 were not conducted.
Groups:
- Placebo: Participants with HCV infection received placebo once daily for 3 days under fasted conditions. This arm was part of cohorts 1, 2 and 3.
- Voxilaprevir 50 mg: Participants with HCV infection received voxilaprevir 50 mg once daily for 3 days under fasted conditions. This arm was part of cohorts 1 and 2.
- Voxilaprevir 100 mg: Participants with HCV infection received voxilaprevir 100 mg once daily for 3 days under fasted conditions. This arm was part of cohorts 1, 2, 3, 4, 5 and 6.
- Voxilaprevir 300 mg: Participants with HCV infection received voxilaprevir 300 mg once daily for 3 days under fasted conditions. This arm was part of cohorts 1 and 2.
- Voxilaprevir 100 mg Fed: Participants with HCV infection received voxilaprevir 100 mg once daily for 3 days under fed conditions. This arm was part of cohorts 1, 2, 3, 4, 5 and 6.
- Voxilaprevir 100 mg + SOF/VEL 400/100 mg: Participants with HCV infection received voxilaprevir 100 mg on Day 1 and voxilaprevir 100 mg plus sofosbuvir (SOF)/velpatasvir (VEL) (400/100 mg) fixed-dose combination (FDC) on Days 2 and 3 after moderate fat or light meal. This arm was part of cohort 10.
Period: Overall Study
Arm/Group | Placebo | Voxilaprevir 50 mg | Voxilaprevir 100 mg | Voxilaprevir 300 mg | Voxilaprevir 100 mg Fed | Voxilaprevir 100 mg + SOF/VEL 400/100 mg
Started | 9 | 20 | 33 | 16 | 7 | 16
Completed | 4 | 7 | 17 | 8 | 4 | 0
Not Completed | 5 | 13 | 16 | 8 | 3 | 16
Not completed — Enrolled but Never Dosed | 1 | 6 | 3 | 1 | 1 | 0
Not completed — Investigator's Discretion | 1 | 0 | 1 | 2 | 2 | 15
Not completed — Withdrew Consent | 2 | 5 | 10 | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 2 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug (voxilaprevir or placebo).
Groups:
- Voxilaprevir 100 mg + SOF/VEL 400/100 mg: Participants with HCV infection received voxilaprevir 100 mg on Day 1 and voxilaprevir 100 mg plus SOF/VEL (400/100 mg) FDC on Days 2 and 3 after moderate fat meal. This arm was part of cohort 10.
- Total: Total of all reporting groups
Arm/Group | Placebo | Voxilaprevir 50 mg | Voxilaprevir 100 mg | Voxilaprevir 300 mg | Voxilaprevir 100 mg Fed | Voxilaprevir 100 mg + SOF/VEL 400/100 mg | Total
Number analyzed (Participants) | 8 | 14 | 30 | 15 | 6 | 16 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (6.1) | 49 (7.7) | 52 (8.0) | 43 (9.4) | 51 (6.2) | 56 (5.2) | 51 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 9 | 5 | 2 | 7 | 29
  Male | 7 | 9 | 21 | 10 | 4 | 9 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 4 | 12 | 3 | 1 | 0 | 22
  White | 6 | 10 | 18 | 12 | 5 | 16 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 12 | 8 | 6 | 9 | 44
  Not Hispanic or Latino | 6 | 7 | 18 | 7 | 0 | 7 | 45
HCV Genotype [Count of Participants; unit: Participants]
  1a | 4 | 8 | 8 | 8 | 0 | 9 | 37
  1b | 0 | 0 | 6 | 0 | 0 | 3 | 9
  2 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  2a/2c | 0 | 0 | 2 | 0 | 0 | 0 | 2
  2b | 2 | 0 | 4 | 0 | 0 | 2 | 8
  3a | 2 | 6 | 6 | 7 | 6 | 1 | 28
  4 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  4a/4c/4d | 0 | 0 | 2 | 0 | 0 | 0 | 2
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.6 (0.39) | 6.0 (0.64) | 6.4 (0.53) | 6.0 (0.64) | 6.0 (0.87) | 6.2 (0.83) | 6.2 (0.65)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 1 | 7 | 6 | 6 | 4 | 4 | 28
  ≥ 800,000 IU/mL | 7 | 7 | 24 | 9 | 2 | 12 | 61

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment Emergent Adverse Events
Time Frame: First dose date up to Day 3 plus 30 days
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug (voxilaprevir or placebo). Data were summarized by dose.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants with HCV infection received placebo once daily for 3 days under fasted conditions. This arm was part of cohorts 1, 2, and 3.
Arm/Group | Placebo | Voxilaprevir 50 mg | Voxilaprevir 100 mg | Voxilaprevir 300 mg | Voxilaprevir 100 mg Fed | Voxilaprevir 100 mg + SOF/VEL 400/100 mg
Number analyzed (Participants) | 8 | 14 | 30 | 15 | 6 | 16
percentage of participants | 25.0 | 14.3 | 16.7 | 13.3 | 33.3 | 12.5

2. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. The severity of laboratory abnormalities was assessed as Grade 0, 1 (mild), 2 (moderate), 3 (severe), or 4 (potentially life threatening) using the Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. The most severe graded abnormality from all tests was counted for each participant.
Time Frame: First dose date up to Day 3 plus 30 days
Population: Participants in the Safety Analysis Set were analyzed. Data were summarized by dose.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Voxilaprevir 50 mg | Voxilaprevir 100 mg | Voxilaprevir 300 mg | Voxilaprevir 100 mg Fed | Voxilaprevir 100 mg + SOF/VEL 400/100 mg
Number analyzed (Participants) | 8 | 14 | 30 | 15 | 6 | 16
percentage of participants
  Grade 1 | 37.5 | 28.6 | 26.7 | 20.0 | 50.0 | 62.5
  Grade 2 | 25.0 | 28.6 | 33.3 | 13.3 | 0 | 12.5
  Grade 3 | 0 | 14.3 | 10.0 | 26.7 | 33.3 | 0
  Grade 4 | 0 | 0 | 3.3 | 0 | 0 | 0

3. Primary Outcome: Antiviral Activity of Voxilaprevir as Measured by Change From Baseline in Plasma HCV RNA
Description: The outcome measure was assessed to evaluate antiviral activity of voxilaprevir only (cohorts 1 through 6). Data are summarized by treatment/cohort and placebo.
Time Frame: Baseline; Days 4, 5, 6, 7, 8, 10, and Week 48
Population: The Efficacy Analysis Set included all enrolled participants with appropriate genotype who received at least one dose of the study drug (voxilaprevir or placebo) and with at least one on-treatment HCV RNA assessment. Participants in the Efficacy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Groups:
- Placebo (GT 1a, Cohort 1): Participants with genotype (GT) 1a HCV infection received placebo once daily for 3 days under fasted conditions.
- Voxilaprevir 50 mg (GT 1a, Cohort 1): Participants with GT 1a HCV infection received voxilaprevir 50 mg once daily for 3 days under fasted conditions.
- Voxilaprevir 100 mg (GT 1a, Cohort 1): Participants with GT 1a HCV infection received voxilaprevir 100 mg once daily for 3 days under fasted conditions.
- Voxilaprevir 300 mg (GT 1a, Cohort 1): Participants with GT 1a HCV infection received voxilaprevir 300 mg once daily for 3 days under fasted conditions.
- Placebo (GT 3, Cohort 2): Participants with GT 3 HCV infection received placebo once daily for 3 days under fasted conditions.
- Voxilaprevir 50 mg (GT 3, Cohort 2): Participants with GT 3 HCV infection received voxilaprevir 50 mg once daily for 3 days under fasted conditions.
- Voxilaprevir 100 mg (GT 3, Cohort 2): Participants with GT 3 HCV infection received voxilaprevir 100 mg once daily for 3 days under fasted conditions.
- Voxilaprevir 300 mg (GT 3, Cohort 2): Participants with GT 3 HCV infection received voxilaprevir 300 mg once daily for 3 days under fasted conditions.
- Placebo (GT 2, Cohort 3): Participants with GT 2 HCV infection received placebo once daily for 3 days under fasted conditions.
- Voxilaprevir 100 mg (GT 2, Cohort 3): Participants with GT 2 HCV infection received voxilaprevir 100 mg once daily for 3 days under fasted conditions.
- Voxilaprevir 100 mg (GT 4, Cohort 4): Participants with GT 4 HCV infection received voxilaprevir 100 mg once daily for 3 days under fasted conditions.
- Voxilaprevir 100 mg (GT 1b, Cohort 5): Participants with GT 1b HCV infection received voxilaprevir 100 mg once daily for 3 days under fasted conditions.
- Voxilaprevir 100 mg Fed (GT 3a, Cohort 6): Participants with GT 3a HCV infection received voxilaprevir 100 mg once daily for 3 days under fed conditions.
Arm/Group | Placebo (GT 1a, Cohort 1) | Voxilaprevir 50 mg (GT 1a, Cohort 1) | Voxilaprevir 100 mg (GT 1a, Cohort 1) | Voxilaprevir 300 mg (GT 1a, Cohort 1) | Placebo (GT 3, Cohort 2) | Voxilaprevir 50 mg (GT 3, Cohort 2) | Voxilaprevir 100 mg (GT 3, Cohort 2) | Voxilaprevir 300 mg (GT 3, Cohort 2) | Placebo (GT 2, Cohort 3) | Voxilaprevir 100 mg (GT 2, Cohort 3) | Voxilaprevir 100 mg (GT 4, Cohort 4) | Voxilaprevir 100 mg (GT 1b, Cohort 5) | Voxilaprevir 100 mg Fed (GT 3a, Cohort 6)
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 2 | 6 | 6 | 7 | 2 | 6 | 4 | 6 | 6
log10 IU/mL
  Change at Day 4: number analyzed (Participants) | 4 | 7 | 8 | 8 | 2 | 5 | 5 | 7 | 2 | 6 | 4 | 6 | 6
  Change at Day 4 | -0.12 (0.136) | -3.81 (0.516) | -3.97 (0.608) | -3.33 (0.902) | -0.24 (0.813) | -1.47 (0.416) | -3.20 (0.364) | -3.57 (0.483) | 0.00 (0.104) | -3.41 (0.444) | -3.50 (0.677) | -3.57 (0.227) | -3.06 (0.752)
  Change at Day 5: number analyzed (Participants) | 4 | 8 | 8 | 7 | 2 | 6 | 5 | 7 | 2 | 6 | 4 | 6 | 6
  Change at Day 5 | -0.20 (0.519) | -3.58 (1.104) | -4.03 (0.594) | -3.37 (0.894) | -0.17 (0.285) | -1.43 (0.606) | -3.00 (0.470) | -3.28 (0.515) | -0.12 (0.151) | -3.37 (0.480) | -3.61 (0.702) | -3.60 (0.390) | -2.45 (0.664)
  Change at Day 6: number analyzed (Participants) | 4 | 8 | 8 | 7 | 2 | 6 | 5 | 7 | 2 | 6 | 4 | 5 | 6
  Change at Day 6 | -0.21 (0.479) | -3.45 (0.829) | -3.78 (0.710) | -3.47 (0.763) | -0.06 (0.051) | -1.06 (0.632) | -2.52 (0.739) | -3.13 (0.736) | -0.04 (0.139) | -3.22 (0.689) | -3.69 (0.879) | -3.61 (0.601) | -2.04 (0.706)
  Change at Day 7: number analyzed (Participants) | 4 | 8 | 8 | 7 | 2 | 6 | 6 | 7 | 2 | 6 | 4 | 6 | 6
  Change at Day 7 | 0.01 (0.340) | -3.15 (0.973) | -3.88 (0.729) | -3.48 (0.695) | 0.02 (0.089) | -0.76 (0.352) | -2.00 (0.378) | -2.89 (0.763) | -0.05 (0.058) | -2.80 (0.494) | -3.70 (0.877) | -3.42 (0.710) | -1.74 (0.885)
  Change at Day 8: number analyzed (Participants) | 4 | 8 | 8 | 7 | 2 | 6 | 5 | 7 | 2 | 6 | 4 | 6 | 6
  Change at Day 8 | 0.13 (0.260) | -2.92 (1.069) | -3.54 (0.663) | -3.23 (0.726) | -0.14 (0.158) | -0.53 (0.379) | -1.79 (0.627) | -2.74 (0.916) | -0.05 (0.090) | -2.48 (0.355) | -3.53 (0.637) | -3.27 (0.627) | -1.43 (0.987)
  Change at Day 10: number analyzed (Participants) | 4 | 8 | 8 | 7 | 2 | 5 | 5 | 7 | 2 | 6 | 4 | 6 | 6
  Change at Day 10 | -0.06 (0.091) | -2.69 (1.116) | -3.33 (0.756) | -2.97 (0.918) | -0.23 (0.180) | -0.28 (0.330) | -1.18 (1.055) | -2.17 (1.394) | -0.13 (0.022) | -2.28 (0.469) | -3.61 (0.674) | -3.08 (0.740) | -0.62 (1.085)
  Change at Week 48: number analyzed (Participants) | 2 | 4 | 7 | 6 | 1 | 3 | 1 | 2 | 1 | 1 | 4 | 5 | 4
  Change at Week 48 | 0.41 (0.873) | 0.08 (0.337) | -0.80 (2.094) | -0.73 (2.352) | 0.41 | -0.03 (0.221) | 0.54 | 0.06 (0.370) | -0.02 | -0.02 | 0.18 (0.247) | -0.57 (2.389) | 0.16 (0.044)

4. Secondary Outcome: Antiviral Activity of Voxilaprevir as Measured by Absolute HCV RNA Level Through Week 48
Description: The outcome measure was assessed to evaluate antiviral activity of voxilaprevir only (cohorts 1 through 6).
Time Frame: Baseline (Pre Day 1 Dose); Days 4, 5, 6, 7, 8, 10, and Week 48
Population: Participants in the Efficacy Analysis Set with available data were analyzed. Data are summarized by treatment/cohort and placebo.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Groups:
- Placebo (GT 1a, Cohort 1): Participants with GT 1a HCV infection received placebo once daily for 3 days under fasted conditions.
Arm/Group | Placebo (GT 1a, Cohort 1) | Voxilaprevir 50 mg (GT 1a, Cohort 1) | Voxilaprevir 100 mg (GT 1a, Cohort 1) | Voxilaprevir 300 mg (GT 1a, Cohort 1) | Placebo (GT 3, Cohort 2) | Voxilaprevir 50 mg (GT 3, Cohort 2) | Voxilaprevir 100 mg (GT 3, Cohort 2) | Voxilaprevir 300 mg (GT 3, Cohort 2) | Placebo (GT 2, Cohort 3) | Voxilaprevir 100 mg (GT 2, Cohort 3) | Voxilaprevir 100 mg (GT 4, Cohort 4) | Voxilaprevir 100 mg (GT 1b, Cohort 5) | Voxilaprevir 100 mg Fed (GT 3a, Cohort 6)
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 2 | 6 | 6 | 7 | 2 | 6 | 4 | 6 | 6
log10 IU/mL
  Pre Day 1 Dose | 6.73 (0.307) | 6.30 (0.497) | 6.35 (0.526) | 6.05 (0.558) | 6.11 (0.480) | 5.61 (0.612) | 6.75 (0.346) | 6.01 (0.773) | 6.71 (0.059) | 6.24 (0.394) | 6.16 (0.730) | 6.23 (0.608) | 6.01 (0.866)
  Day 4: number analyzed (Participants) | 4 | 7 | 8 | 8 | 2 | 5 | 5 | 7 | 2 | 6 | 4 | 6 | 6
  Day 4 | 6.62 (0.378) | 2.56 (0.705) | 2.38 (0.759) | 2.72 (0.943) | 5.87 (0.332) | 4.22 (0.878) | 3.54 (0.455) | 2.44 (0.693) | 6.71 (0.164) | 2.83 (0.611) | 2.65 (0.533) | 2.67 (0.500) | 2.95 (0.505)
  Day 5: number analyzed (Participants) | 4 | 8 | 8 | 7 | 2 | 6 | 5 | 7 | 2 | 6 | 4 | 6 | 6
  Day 5 | 6.53 (0.426) | 2.73 (1.203) | 2.33 (0.643) | 2.67 (0.947) | 5.94 (0.195) | 4.19 (1.104) | 3.75 (0.455) | 2.73 (0.780) | 6.59 (0.210) | 2.87 (0.603) | 2.55 (0.549) | 2.63 (0.764) | 3.56 (0.273)
  Day 6: number analyzed (Participants) | 4 | 8 | 8 | 7 | 2 | 6 | 5 | 7 | 2 | 6 | 4 | 5 | 6
  Day 6 | 6.52 (0.320) | 2.85 (1.000) | 2.57 (1.028) | 2.57 (0.818) | 6.05 (0.532) | 4.55 (1.203) | 4.23 (0.604) | 2.88 (0.882) | 6.68 (0.199) | 3.02 (0.754) | 2.46 (0.300) | 2.85 (0.685) | 3.98 (0.413)
  Day 7: number analyzed (Participants) | 4 | 8 | 8 | 7 | 2 | 6 | 5 | 7 | 2 | 6 | 4 | 6 | 6
  Day 7 | 6.74 (0.059) | 3.15 (1.268) | 2.47 (0.821) | 2.56 (0.714) | 6.13 (0.569) | 4.85 (0.886) | 4.75 (0.268) | 3.12 (0.991) | 6.67 (0.001) | 3.44 (0.613) | 2.45 (0.359) | 2.82 (1.111) | 4.27 (0.485)
  Day 8: number analyzed (Participants) | 4 | 8 | 8 | 7 | 2 | 6 | 5 | 7 | 2 | 6 | 4 | 6 | 6
  Day 8 | 6.86 (0.144) | 3.38 (1.019) | 2.81 (0.901) | 2.81 (0.671) | 5.97 (0.323) | 5.08 (0.655) | 4.96 (0.531) | 3.27 (1.100) | 6.66 (0.031) | 3.76 (0.497) | 2.62 (0.278) | 2.96 (1.111) | 4.59 (0.528)
  Day 10: number analyzed (Participants) | 4 | 8 | 8 | 7 | 2 | 5 | 5 | 7 | 2 | 6 | 4 | 6 | 6
  Day 10 | 6.68 (0.263) | 3.61 (1.041) | 3.03 (0.857) | 3.07 (0.887) | 5.88 (0.300) | 5.43 (0.803) | 5.56 (0.987) | 3.83 (1.417) | 6.58 (0.081) | 3.96 (0.555) | 2.54 (0.553) | 3.15 (1.210) | 5.40 (0.697)
  Week 48: number analyzed (Participants) | 2 | 4 | 7 | 6 | 1 | 3 | 1 | 2 | 1 | 1 | 4 | 5 | 4
  Week 48 | 6.97 (0.488) | 6.29 (0.825) | 5.55 (2.007) | 5.20 (2.085) | 6.18 | 5.13 (0.207) | 7.29 | 6.38 (1.479) | 6.65 | 6.13 | 6.34 (0.696) | 5.65 (2.473) | 5.98 (0.891)

5. Secondary Outcome: Antiviral Activity of Voxilaprevir as Measured by Number of Participants Achieving Reductions From Baseline in HCV RNA
Description: Categorical declines from baseline were summarized by the number of participants with a < 1, ≥ 1 to <2, ≥ 2 to <3, or ≥ 3 log10 IU/mL decrease in HCV RNA from baseline to each postdose assessment up to Week 48 by treatment/cohort and placebo. The outcome measure was assessed to evaluate antiviral activity of voxilaprevir only (cohorts 1 through 6).
Time Frame: Baseline; Days 4, 5, 6, 7, 8, 10, and Week 48
Population: Participants in the Efficacy Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (GT 1a, Cohort 1) | Voxilaprevir 50 mg (GT 1a, Cohort 1) | Voxilaprevir 100 mg (GT 1a, Cohort 1) | Voxilaprevir 300 mg (GT 1a, Cohort 1) | Placebo (GT 3, Cohort 2) | Voxilaprevir 50 mg (GT 3, Cohort 2) | Voxilaprevir 100 mg (GT 3, Cohort 2) | Voxilaprevir 300 mg (GT 3, Cohort 2) | Placebo (GT 2, Cohort 3) | Voxilaprevir 100 mg (GT 2, Cohort 3) | Voxilaprevir 100 mg (GT 4, Cohort 4) | Voxilaprevir 100 mg (GT 1b, Cohort 5) | Voxilaprevir 100 mg Fed (GT 3a, Cohort 6)
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 2 | 6 | 6 | 7 | 2 | 6 | 4 | 6 | 6
Participants
  Day 4: Missing HCV RNA | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 4: < 1 log10 IU/mL decrease in HCV RNA | 4 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Day 4: ≥1 and <2 log10 IU/mL decrease in HCV RNA | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 4: ≥2 and <3 log10 IU/mL decrease in HCV RNA | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 3
  Day 4: ≥3 log10 IU/mL decrease in HCV RNA | 0 | 7 | 7 | 7 | 0 | 0 | 4 | 6 | 0 | 5 | 3 | 6 | 3
  Day 5: Missing HCV RNA | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 5: < 1 log10 IU/mL decrease in HCV RNA | 4 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Day 5: ≥1 and <2 log10 IU/mL decrease in HCV RNA | 0 | 1 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Day 5: ≥2 and <3 log10 IU/mL decrease in HCV RNA | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 2 | 1 | 0 | 3
  Day 5: ≥3 log10 IU/mL decrease in HCV RNA | 0 | 6 | 8 | 6 | 0 | 0 | 3 | 5 | 0 | 4 | 3 | 6 | 2
  Day 6: Missing HCV RNA | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Day 6: < 1 log10 IU/mL decrease in HCV RNA | 4 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Day 6: ≥1 and <2 log10 IU/mL decrease in HCV RNA | 0 | 1 | 0 | 1 | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 3
  Day 6: ≥2 and <3 log10 IU/mL decrease in HCV RNA | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 1 | 1 | 2
  Day 6: ≥3 log10 IU/mL decrease in HCV RNA | 0 | 7 | 7 | 6 | 0 | 0 | 1 | 5 | 0 | 4 | 3 | 4 | 1
  Day 7: Missing HCV RNA | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 7: < 1 log10 IU/mL decrease in HCV RNA | 4 | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 2 | 0 | 0 | 0 | 1
  Day 7: ≥1 and <2 log10 IU/mL decrease in HCV RNA | 0 | 2 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 2
  Day 7: ≥2 and <3 log10 IU/mL decrease in HCV RNA | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 3 | 1 | 2 | 3
  Day 7: ≥3 log10 IU/mL decrease in HCV RNA | 0 | 6 | 7 | 6 | 0 | 0 | 0 | 4 | 0 | 3 | 3 | 4 | 0
  Day 8: Missing HCV RNA | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8: < 1 log10 IU/mL decrease in HCV RNA | 4 | 0 | 0 | 0 | 2 | 6 | 0 | 1 | 2 | 0 | 0 | 0 | 3
  Day 8: ≥1 and <2 log10 IU/mL decrease in HCV RNA | 0 | 2 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 2
  Day 8: ≥2 and <3 log10 IU/mL decrease in HCV RNA | 0 | 2 | 1 | 3 | 0 | 0 | 1 | 2 | 0 | 6 | 1 | 2 | 1
  Day 8: ≥3 log10 IU/mL decrease in HCV RNA | 0 | 4 | 7 | 4 | 0 | 0 | 0 | 4 | 0 | 0 | 3 | 4 | 0
  Day 10: Missing HCV RNA | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 10: < 1 log10 IU/mL decrease in HCV RNA | 4 | 0 | 0 | 0 | 2 | 5 | 2 | 1 | 2 | 0 | 0 | 0 | 4
  Day 10: ≥1 and <2 log10 IU/mL decrease in HCV RNA | 0 | 3 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 1 | 1
  Day 10: ≥2 and <3 log10 IU/mL decrease in HCV RNA | 0 | 2 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 4 | 0 | 1 | 1
  Day 10: ≥3 log10 IU/mL decrease in HCV RNA | 0 | 3 | 7 | 3 | 0 | 0 | 0 | 3 | 0 | 0 | 4 | 4 | 0
  Week 48: Missing HCV RNA | 2 | 4 | 1 | 2 | 1 | 3 | 5 | 5 | 1 | 5 | 0 | 1 | 2
  Week 48: < 1 log10 IU/mL decrease in HCV RNA | 2 | 4 | 6 | 5 | 1 | 3 | 1 | 2 | 1 | 1 | 4 | 4 | 4
  Week 48: ≥1 and <2 log10 IU/mL decrease in HCV RNA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 48: ≥2 and <3 log10 IU/mL decrease in HCV RNA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 48: ≥3 log10 IU/mL decrease in HCV RNA | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

6. Secondary Outcome: Percentage of Participants Who Have HCV RNA < Lower Limit of Quantitation (LLOQ) Detected, and < LLOQ Target Not Detected (TND)
Description: The lower limit of quantitation (LLOQ) detection for HCV RNA levels was 15 IU/mL. HCV detected means calculated HCV RNA level is below LLOQ of the assay. The outcome measure was assessed to evaluate antiviral activity of voxilaprevir only (cohorts 1 through 6).
Time Frame: Days 4, 5, 6, 7, 8, 10, and Week 48
Population: Participants in the Efficacy Analysis Set were analyzed. Data are summarized by treatment/cohort and placebo.
Measure: Number; unit: participants
Arm/Group | Placebo (GT 1a, Cohort 1) | Voxilaprevir 50 mg (GT 1a, Cohort 1) | Voxilaprevir 100 mg (GT 1a, Cohort 1) | Voxilaprevir 300 mg (GT 1a, Cohort 1) | Placebo (GT 3, Cohort 2) | Voxilaprevir 50 mg (GT 3, Cohort 2) | Voxilaprevir 100 mg (GT 3, Cohort 2) | Voxilaprevir 300 mg (GT 3, Cohort 2) | Placebo (GT 2, Cohort 3) | Voxilaprevir 100 mg (GT 2, Cohort 3) | Voxilaprevir 100 mg (GT 4, Cohort 4) | Voxilaprevir 100 mg (GT 1b, Cohort 5) | Voxilaprevir 100 mg Fed (GT 3a, Cohort 6)
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 2 | 6 | 6 | 7 | 2 | 6 | 4 | 6 | 6
participants
  Day 4 < LLOQ detected | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 5 < LLOQ detected | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Day 6 < LLOQ TND | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 7 < LLOQ detected | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Day 8 < LLOQ detected | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Day 10 < LLOQ TND | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 48 < LLOQ TND | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to Day 3 plus 30 days; All-Cause Mortality: First dose date up to Week 48
Description: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug (voxilaprevir or placebo). Data were summarized by dose.
Arm/Group | Placebo | Voxilaprevir 50 mg | Voxilaprevir 100 mg | Voxilaprevir 300 mg | Voxilaprevir 100 mg Fed | Voxilaprevir 100 mg + SOF/VEL 400/100 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/14 | 0/30 | 0/15 | 0/6 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/14 | 0/30 | 0/15 | 1/6 | 0/16
Other Adverse Events (participants affected / at risk) | 2/8 | 2/14 | 2/30 | 2/15 | 1/6 | 2/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | Voxilaprevir 50 mg (N=14) | Voxilaprevir 100 mg (N=30) | Voxilaprevir 300 mg (N=15) | Voxilaprevir 100 mg Fed (N=6) | Voxilaprevir 100 mg + SOF/VEL 400/100 mg (N=16)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | Voxilaprevir 50 mg (N=14) | Voxilaprevir 100 mg (N=30) | Voxilaprevir 300 mg (N=15) | Voxilaprevir 100 mg Fed (N=6) | Voxilaprevir 100 mg + SOF/VEL 400/100 mg (N=16)
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 1 | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years